CLINICAL TRIAL: NCT00732069
Title: Genes, Fibrinolysis and Endothelial Dysfunction- Dialysis Aim 2
Brief Title: Study of Inflammation and Oxidative Stress in Persons Undergoing Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nancy J. Brown, Professor, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fibrinolysis in Dialysis; R01HL065193-08A2 (NIH)
Record Dates: First submitted 2008-08-06; First posted 2008-08-11 (Estimated); Results first posted 2013-06-20 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: End Stage Renal Failure on Dialysis; Complication of Hemodialysis
Keywords: hemodialysis; oxidative stress; inflammation; kallikrein-kinin; angiotensin receptor blockade; angiotensin converting enzyme inhibition; RAAS; fibrinolysis; endothelial dysfunction
MeSH Terms: conditions — Inflammation | interventions — Ramipril; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo, then ramipril, then valsartan (Active Comparator): placebo, ramipril, valsartan: Subjects were treated sequentially with placebo, ramipril (5mg/day by mouth), then valsartan (160mg/day by mouth). Each drug was given for 7 days after a 3-week washout.
  Interventions: Drug: Placebo; Drug: Ramipril; Drug: Valsartan
- Placebo, then valsartan, then ramipril (Active Comparator): placebo, ramipril, valsartan: Subjects were treated sequentially with placebo, valsartan (160mg/day by mouth), then ramipril (5mg/day by mouth). Each drug was given for 7 days after a 3-week washout.
  Interventions: Drug: Placebo; Drug: Ramipril; Drug: Valsartan
- Ramipril, then placebo, then valsartan (Active Comparator): placebo, ramipril, valsartan: Subjects were treated sequentially with ramipril (5mg/day by mouth), then placebo (once a day by mouth), then valsartan (160mg/day by mouth). Each drug was given for 7 days after a 3-week washout.
  Interventions: Drug: Placebo; Drug: Ramipril; Drug: Valsartan
- Valsartan, then placebo, then ramipril (Active Comparator): placebo, ramipril, valsartan: Subjects were treated sequentially with valsartan (160mg/day by mouth), then placebo (once a day by mouth), then ramipril (5mg/day by mouth). Each drug was given for 7 days after a 3-week washout.
  Interventions: Drug: Placebo; Drug: Ramipril; Drug: Valsartan
- Ramipril, then valsartan, then placebo (Active Comparator): placebo, ramipril, valsartan: Subjects were treated sequentially with ramipril (5mg/day by mouth), then valsartan (160mg/day by mouth), then placebo (once a day by mouth). Each drug was given for 7 days after a 3-week washout.
  Interventions: Drug: Placebo; Drug: Ramipril; Drug: Valsartan
- Valsartan, then ramipril, then placebo (Active Comparator): placebo, ramipril, valsartan: Subjects were treated sequentially with then valsartan (160mg/day by mouth), then ramipril (5mg/day by mouth), then placebo (once a day by mouth). Each drug was given for 7 days after a 3-week washout.
  Interventions: Drug: Placebo; Drug: Ramipril; Drug: Valsartan

INTERVENTIONS:
Drug: Placebo — Patients receiving an angiotensin converting enzyme inhibitor or angiotensin receptor blocker before the study underwent washout for 3 weeks. Subjects were treated with study drug for 7 days and each treatment period was separated by a 3-week washout period. Ramipril was given at dose of 2.5mg/d for two days, then 5mg/d for 5 days. Valsartan was given at 80mg/d for 2 days followed by 160mg/d for 5 days. On the seventh day of each treatment blood samples were collected prior two, during and two hours after dialysis
  Other Names: matching placebo
Drug: Ramipril — Patients receiving an angiotensin converting enzyme inhibitor or angiotensin receptor blocker before the study underwent washout for 3 weeks. Subjects were treated with study drug for 7 days and each treatment period was separated by a 3-week washout period. Ramipril was given at dose of 2.5mg/d for two days, then 5mg/d for 5 days. Valsartan was given at 80mg/d for 2 days followed by 160mg/d for 5 days. On the seventh day of each treatment blood samples were collected prior two, during and two hours after dialysis
  Other Names: Ramipril 2.5mg/d for two days, then 5mg/d for 5 days.
Drug: Valsartan — Patients receiving an angiotensin converting enzyme inhibitor or angiotensin receptor blocker before the study underwent washout for 3 weeks. Subjects were treated with study drug for 7 days and each treatment period was separated by a 3-week washout period. Ramipril was given at dose of 2.5mg/d for two days, then 5mg/d for 5 days. Valsartan was given at 80mg/d for 2 days followed by 160mg/d for 5 days. On the seventh day of each treatment blood samples were collected prior two, during and two hours after dialysis
  Other Names: Valsartan 80mg/d for 2 days followed by 160mg/d for 5 days.

SUMMARY:
Little is known about how some drugs affect inflammation or clotting factors in people receiving hemodialysis. It is not yet known if these drugs help prevent heart damage as they do in people not undergoing hemodialysis or whether they could increase the risk of heart problems. The purpose of the study is to measure certain chemicals in the blood and see how those chemicals may change during hemodialysis when certain drugs are given.

DETAILED DESCRIPTION:
* Cardiovascular disease in the leading cause of death in patients with chronic kidney disease undergoing hemodialysis.
* Traditional risk factors do not adequately predict cardiovascular morbidity and mortality in patients with chronic kidney disease.
* Increased oxidative stress, inflammation and impaired fibrinolysis contribute to cardiovascular risk in chronic kidney disease patients undergoing hemodialysis.
* Activation of the renin-angiotensin-aldosterone system(RAAS) may contribute to oxidative stress and inflammation in individuals with chronic kidney disease
* Activation of the kallikrein-kinin system during hemodialysis may increase fibrinolysis but may also contribute to inflammation in chronic kidney disease
* Despite data from clinical trials demonstrating that ARBs and ACE inhibitors decrease cardiovascular mortality, delay progression to cardiovascular disease and decrease the incidence of diabetes in the general population little is known about the impact of these agents on cardiovascular morbidity and mortality in patients with end- stage renal disease (ESRD) undergoing hemodialysis
* Angiotensin-converting enzyme(ACE) inhibitors and angiotensin receptor blockers (ARB)S differ in their mechanisms of action and their effects on inflammatory biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* On thrice-weekly chronic hemodialysis for at least 6 months
* Clinically stable, adequately dialyzed (single-pool Kt/V> 1.2) thrice weekly, with polysulphone membrane for at least 3 consecutive months prior to study

Exclusion Criteria:

* Body mass index > 35 mg/kg
* History of functional transplant less than 6 months prior to study
* Use of anti-inflammatory medications other than aspirin < 325 mg/d
* History of active connective tissue disease
* History of acute infectious disease within one month prior to study
* AIDS (HIV seropositivity is not an exclusion criteria)
* History of myocardial infarction or cerebrovascular event within 3 months
* Advanced liver disease
* Gastrointestinal dysfunction requiring parental nutrition
* Active malignancy excluding basal cell carcinoma of the skin
* History of ACE inhibitor-associated cough or angioedema
* Ejection fraction less than 40%
* Inability to discontinue ACE inhibitor or ARB
* Predialysis potassium repeatedly higher than 5.5 mmol/L (confirmed on a repeated blood draw)
* Anticipated live donor kidney transplant
* Use of vitamin E >60 IU/d or vitamin C >500 mg/d
* Pregnancy, breast-feeding or child-bearing potential
* History of poor adherence to hemodialysis or medical regimen
* Inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Gamboa JL, Pretorius M, Todd-Tzanetos DR, Luther JM, Yu C, Ikizler TA, Brown NJ. Comparative effects of angiotensin-converting enzyme inhibition and angiotensin-receptor blockade on inflammation during hemodialysis. J Am Soc Nephrol. 2012 Feb;23(2):334-42. doi: 10.1681/ASN.2011030287. Epub 2011 Dec 8. PMID 22158433
- [Derived] Gamboa JL, Pretorius M, Sprinkel KC, Brown NJ, Ikizler TA. Angiotensin converting enzyme inhibition increases ADMA concentration in patients on maintenance hemodialysis--a randomized cross-over study. BMC Nephrol. 2015 Oct 22;16:167. doi: 10.1186/s12882-015-0162-x. PMID 26494370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in September 2008 and ended in January 2010 in Vanderbilt outpatients Dialysis Center.
Pre-assignment Details: Three consented participants were excluded because of hyperkalemia, hypotension and uncontrollable hypertension.They were enrolled but did not start medication and were considered screen failures. The participants required a washout period from either an agiotensin receptor blocker or an angiotensin converting enzyme inhibitor.
Groups:
- Placebo, Then Ramipril, Then Valsartan; Placebo, Valsartan, Then Ramipril; Ramipril, Then Placebo, Then Valsartan; Valsartan, Then Placebo, Then Ramipril; Ramipril, Valsartan, Then Placebo; Valsartan, Ramipril, Then Placebo: Participants were randomized to treatment with ramipril, valsartan and placebo in one of six possible sequences.
Period: First Study Drug
Arm/Group | Placebo, Then Ramipril, Then Valsartan | Placebo, Valsartan, Then Ramipril | Ramipril, Then Placebo, Then Valsartan | Valsartan, Then Placebo, Then Ramipril | Ramipril, Valsartan, Then Placebo | Valsartan, Ramipril, Then Placebo
Started | 3 | 3 | 3 | 2 | 3 | 2
Completed | 3 | 3 | 3 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout After First Study Drug
Arm/Group | Placebo, Then Ramipril, Then Valsartan | Placebo, Valsartan, Then Ramipril | Ramipril, Then Placebo, Then Valsartan | Valsartan, Then Placebo, Then Ramipril | Ramipril, Valsartan, Then Placebo | Valsartan, Ramipril, Then Placebo
Started | 3 | 3 | 3 | 2 | 3 | 2
Completed | 2 | 3 | 3 | 2 | 3 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Second Study Drug
Arm/Group | Placebo, Then Ramipril, Then Valsartan | Placebo, Valsartan, Then Ramipril | Ramipril, Then Placebo, Then Valsartan | Valsartan, Then Placebo, Then Ramipril | Ramipril, Valsartan, Then Placebo | Valsartan, Ramipril, Then Placebo
Started | 2 | 3 | 3 | 2 | 3 | 2
Completed | 2 | 3 | 3 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout After Second Study Drug
Arm/Group | Placebo, Then Ramipril, Then Valsartan | Placebo, Valsartan, Then Ramipril | Ramipril, Then Placebo, Then Valsartan | Valsartan, Then Placebo, Then Ramipril | Ramipril, Valsartan, Then Placebo | Valsartan, Ramipril, Then Placebo
Started | 2 | 3 | 3 | 2 | 3 | 2
Completed | 2 | 3 | 3 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Study Drug
Arm/Group | Placebo, Then Ramipril, Then Valsartan | Placebo, Valsartan, Then Ramipril | Ramipril, Then Placebo, Then Valsartan | Valsartan, Then Placebo, Then Ramipril | Ramipril, Valsartan, Then Placebo | Valsartan, Ramipril, Then Placebo
Started | 2 | 3 | 3 | 2 | 3 | 2
Completed | 2 | 3 | 3 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: After a three week washout period, the subject will be undertake 3 study periods with one of three treatments, placebo, ramipril or valsartan
Arm/Group | All Study Participants
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 50.5 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Interleukin 1 Beta
Description: Mean difference in interleukin 1 beta concentration during treatment with ramipril versus treatment with placebo
Time Frame: During dialysis after one week of study drug
Population: All participants who completed the three arm treatment.
Measure: Mean (Standard Error); unit: pg/mL
Groups:
- Ramipril; Valsartan; Placebo: After a three week washout period, the subject will be undertake 3 study periods with one of three treatments, placebo, ramipril or valsartan
Arm/Group | Ramipril | Valsartan | Placebo
Number analyzed (Participants) | 15 | 15 | 15
pg/mL | 6.18 (3.56) | 2.16 (2.16) | 1.44 (1.49)

2. Secondary Outcome: F2-Isoprostanes
Description: Mean difference in F2-isoprostanes during dialysis between treatment with ramipril or valsartan and placebo
Time Frame: During dialysis after one week of study drug
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ramipril | Valsartan | Placebo
Number analyzed (Participants) | 15 | 15 | 15
pg/mL | 59.55 (27.53) | 59.03 (29.39) | 50.23 (22.59)

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Ramipril: All subjects receiving ramipril
- Valsartan: All subjects receiving valsartan
- Placebo: All subjects receiving placebo
Arm/Group | Ramipril | Valsartan | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 1/16
Other Adverse Events (participants affected / at risk) | 1/15 | 4/15 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramipril (N=15) | Valsartan (N=15) | Placebo (N=16)
Cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Patient develop acute occipital infarct without evidence of hemorrhage within the 3 weeks washout period after receiving placebo treatment. The stroke was not felt to be study related by the Data and Safety Monitoring Committee for this study
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramipril (N=15) | Valsartan (N=15) | Placebo (N=15)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) — Both episodes of nausea occurred during valsartan treatment.
Hypotension (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) — One event each during ramipril, valsartan, placebo treatment
Dry cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Occurred during placebo
Chest pain not cardiac (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Event occurred during placebo
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Occurred during placebo
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) — 1 event during valsartan, one in a subject during placebo
Bruising after falling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Occurred in subject taking placebo
Vascular acces complication (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — occurred during placebo

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No